CLINICAL TRIAL: NCT03847753
Title: Exploring the Comorbidity Between Mental Disorders and General Medical Conditions Among a Danish National Population
Brief Title: Exploring the Comorbidity Between Mental Disorders and General Medical Conditions
Acronym: COMO-GMC
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: COMO-GMC
Record Dates: First submitted 2019-02-07; First posted 2019-02-20 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-04

CONDITIONS: Organic, Including Symptomatic, Mental Disorders; Substance Use; Schizophrenia; Mood [Affective] Disorders; Neurotic, Stress-related and Somatoform Disorders; Eating Disorder; Disorders of Adult Personality and Behavior; Mental Retardation; Disorder of Psychological Development; Behavioural Disorder; Hypertension; Dyslipidemias; Ischemic Heart Disease; Atrial Fibrillation; Heart Failure; Peripheral Occlusive Disease; Stroke; Diabetes Mellitus; Thyroid Disorder; Gout; Chronic Pulmonary Disease; Allergy; Chronic Gastritis; Chronic Liver Disease; Inflammatory Bowel Diseases; Diverticular Disease of Large Intestine; Chronic Kidney Diseases; Prostate Disorders; Connective Tissue Disorder; Osteoporosis; Pain; HIV/AIDS; Anemia; Cancer; Vision Disorders; Hearing Disorders; Migraine; Epilepsy; Parkinson Disease; Multiple Sclerosis; Neuropathy
Keywords: Comorbidity
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Schizophrenia; Mood Disorders; Somatoform Disorders; Feeding and Eating Disorders; Behavior; Intellectual Disability; Hypertension; Dyslipidemias; Myocardial Ischemia; Atrial Fibrillation; Heart Failure; Stroke; Diabetes Mellitus; Thyroid Diseases; Gout; Hypersensitivity; Inflammatory Bowel Diseases; Renal Insufficiency, Chronic; Prostatic Diseases; Connective Tissue Diseases; Osteoporosis; Pain; Acquired Immunodeficiency Syndrome; Anemia; Neoplasms; Vision Disorders; Hearing Disorders; Migraine Disorders; Epilepsy; Parkinson Disease; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 17 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Danish population: The cohort includes all those born in Denmark between 1900-2015, and who resided there in the period of 2000-2016.Whether they received a diagnosis of one of the following mental disorders will be ascertained: Organic Disorders, Substance Use Disorders, Schizophrenia Disorders, Mood Disorders, Eating Disorders, Neurotic Disorders, Personality Disorders, Intellectual Disorders, Developmental Disorders, Behavioral Disorders The risk of receiving a later diagnosis of one of the following types of general medical conditions will then be estimated: Circulatory, Endocrine, Pulmonary and Allergy, Gastrointestinal, Urogenital, Musculoskeletal, Hematological, Cancer, Neurological
  Interventions: Other: Organic Disorders; Other: Substance Use Disorders; Other: Schizophrenia Disorders; Other: Mood disorders; Other: Neurotic disorders; Other: Eating Disorders; Other: Personality Disorders; Other: Intellectual Disorders; Other: Developmental Disorders; Other: Behavioral Disorders

INTERVENTIONS:
Other: Organic Disorders — Individuals were considered to have a specific mental disorder from the date they received a relevant diagnosis registered in the Danish Psychiatric Central Research Register.
Other: Substance Use Disorders — Individuals were considered to have a specific mental disorder from the date they received a relevant diagnosis registered in the Danish Psychiatric Central Research Register.
Other: Schizophrenia Disorders — Individuals were considered to have a specific mental disorder from the date they received a relevant diagnosis registered in the Danish Psychiatric Central Research Register.
Other: Mood disorders — Individuals were considered to have a specific mental disorder from the date they received a relevant diagnosis registered in the Danish Psychiatric Central Research Register.
Other: Neurotic disorders — Individuals were considered to have a specific mental disorder from the date they received a relevant diagnosis registered in the Danish Psychiatric Central Research Register.
Other: Eating Disorders — Individuals were considered to have a specific mental disorder from the date they received a relevant diagnosis registered in the Danish Psychiatric Central Research Register.
Other: Personality Disorders — Individuals were considered to have a specific mental disorder from the date they received a relevant diagnosis registered in the Danish Psychiatric Central Research Register.
Other: Intellectual Disorders — Individuals were considered to have a specific mental disorder from the date they received a relevant diagnosis registered in the Danish Psychiatric Central Research Register.
Other: Developmental Disorders — Individuals were considered to have a specific mental disorder from the date they received a relevant diagnosis registered in the Danish Psychiatric Central Research Register.
Other: Behavioral Disorders — Individuals were considered to have a specific mental disorder from the date they received a relevant diagnosis registered in the Danish Psychiatric Central Research Register.

SUMMARY:
Mental disorders have been shown to be associated with a number of general medical conditions (also referred to as somatic or physical conditions). The investigators aim to undertake a comprehensive study of comorbidity among those with treated mental disorders, by using high-quality Danish registers to provide age- and sex-specific pairwise estimates between the ten groups of mental disorders and nine groups of general medical conditions.

The investigators will examine the association between all 90 possible pairs of prior mental disorders and later GMC categories using the Danish national registers. Depending on whether individuals are diagnosed with a specific mental disorder, the investigators will estimate the risk of receiving a later diagnosis within a specific GMC category, between the start of follow-up (January 1, 2000) or at the earliest age at which a person might develop the mental disorder, whichever comes later. Follow-up will be terminated at onset of the GMC, death, emigration from Denmark, or December 31, 2016, whichever came first. Additionally for dyslipidemia, follow-up will be ended if a diagnosis of ischemic heart disease was received. A "wash-out" period will be employed in the five years before follow-up started (1995-1999), to identify and exclude prevalent cases from the analysis. Individuals with the GMC of interest before the observation period will be considered prevalent cases and excluded from the analyses (i.e. prevalent cases were "washed-out"). When estimating the risk of a specific GMC, the investigators will consider all individuals to be exposed or unexposed to the each mental disorder depending on whether a diagnosis is received before the end of follow-up. Persons will be considered unexposed to a mental disorder until the date of the first diagnosis, and exposed thereafter.

DETAILED DESCRIPTION:
The investigators will analyse data from all individuals born in Denmark between 1900-2015 and who resided there between 2000-2016; giving a study size of over 5.5 million people. The National Patient Register, Cause of Death Register and National Prescription Registry of Denmark will all be used as sources of information about the mental disorders and general medical conditions (GMC) of interest. These are considered to be of high quality and validity.

The rate of diagnosis with a specific GMC group between those exposed and unexposed to each of ten mental disorders will be examined using hazard ratios (HRs) and 95% confidence intervals (CI), using Cox proportional hazards models with age as the underlying time scale. The following models will be run to provide all persons and sex-specific estimates, considering exposure to each mental disorder and whether the association differs depending on the time since onset of the mental disorder (lagged HRs):

Model A: adjusted for sex and birth date which, in combination with underlying age in the models, adjusts also for calendar time

Model B: additionally adjust for mental disorder comorbidity with onset before, but not after, the mental disorder of interest

Finally, cumulative incidence proportions of diagnosis with a GMC after being diagnosed with a mental disorder will be estimated. This will provide absolute risks of developing a GMC after a specific time, given a previous diagnosis of a mental disorder. To compare cumulative incidence proportions among people diagnosed with a mental disorder to those among people without a diagnosis, a matched reference group will be generated for each mental disorder. For every index person with the mental disorder, up to five age- and sex-matched individuals (who had not received a diagnosis of the relevant mental disorder by the age the index person was diagnosed) will be randomly selected. Cumulative incidence proportions will be generated for each reference group. All analyses will be performed on the secured platform of Statistics Denmark STATA/MP version 15.1 (Stata Corporation, College Station, Texas, USA).

An interactive webpage will be developed to visualize all results from this study. The Danish Data Protection Agency and the Danish Health Data Authority approved this study.

ELIGIBILITY:
Inclusion Criteria:

* Born in Denmark between 1900-2015
* Resided in Denmark during the study period (2000-2016)

Exclusion Criteria:

* Excluded from analyses for each specific GMC, if considered a prevalent case of that GMC (i.e. ascertained to have a diagnosis for the GMC during the washout period of 1995-1999)

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All individuals born in Denmark between 1900-2015 and who resided there between 2000-2016
Sampling Method: Non-Probability Sample
Enrollment: 5940299 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Risk of circulatory system general medical conditions | Diagnosed during the study period (2000-2016), after at least 1 year of age
  These will be ascertained using the following criteria:
  Diagnosis in the Danish National Patient Register or death in the Cause of Death register, for at least one of the following diseases: hypertension, dyslipidemia, ischemic heart disease, atrial fibrillation, heart failure, peripheral arterial occlusive disease, stroke.
  Records in the Danish National Prescription Register for at least one of the following types of medications: antihypertensives, lipid-lowering drugs, antianginal drugs (at least two prescriptions for a type of medication in one year).
  Hazard ratios (HRs), with 95% confidence intervals, will be obtained to compare risk of diagnosis with a general medical condition in those with previous mental disorders, compared to those without. All persons, sex-specific and lagged (accounting for time since mental disorder diagnosis) HRs will be obtained. Additionally absolute risks will be calculated.
Risk of Endocrine System general medical conditions | Diagnosed during the study period (2000-2016), after at least 1 year of age
  These will be ascertained using the following criteria:
  Diagnosis in the Danish National Patient Register or death in the Cause of Death register, for at least one of the following diseases: diabetes mellitus, thyroid disorders, gout.
  Records in the Danish National Prescription Register for at least one of the following types of medications: antidiabetic, thyroid therapy drugs (at least two prescriptions for a type of medication in one year).
  Hazard ratios (HRs), with 95% confidence intervals, will be obtained to compare risk of diagnosis with a general medical condition in those with previous mental disorders, compared to those without. All persons, sex-specific and lagged (accounting for time since mental disorder diagnosis) HRs will be obtained. Additionally absolute risks will be calculated.
Risk of Pulmonary System general medical conditions | Diagnosed during the study period (2000-2016), after at least 1 year of age
  These will be ascertained using the following criteria:
  Diagnosis in the Danish National Patient Register or death in the Cause of Death register, for at least one of the following diseases: chronic pulmonary disease, allergy.
  Records in the Danish National Prescription Register for at least one of the following types of medications: obstructive airway disease drugs, non-sedative antihistamines and/or nasal antiallergics (at least two prescriptions for a type of medication in one year).
  Hazard ratios (HRs), with 95% confidence intervals, will be obtained to compare risk of diagnosis with a general medical condition in those with previous mental disorders, compared to those without. All persons, sex-specific and lagged (accounting for time since mental disorder diagnosis) HRs will be obtained. Additionally absolute risks will be calculated.
Risk of Gastrointestinal System general medical conditions | Diagnosed during the study period (2000-2016), after at least 1 year of age
  These will be ascertained using the following criteria:
  Diagnosis in the Danish National Patient Register or death in the Cause of Death register, for at least one of the following diseases: ulcer/chronic gastritis, chronic liver disease, inflammatory bowel disease, diverticular disease of intestine.
  Hazard ratios (HRs), with 95% confidence intervals, will be obtained to compare risk of diagnosis with a general medical condition in those with previous mental disorders, compared to those without. All persons, sex-specific and lagged (accounting for time since mental disorder diagnosis) HRs will be obtained. Additionally absolute risks will be calculated.
Risk of Urogenital System general medical conditions | Diagnosed during the study period (2000-2016), after at least 1 year of age
  These will be ascertained using the following criteria:
  Diagnosis in the Danish National Patient Register or death in the Cause of Death register, for at least one of the following diseases: chronic kidney disease, prostate disorders.
  Records in the Danish National Prescription Register for at least one of the following types of medications: prostate hyperplasia therapy drugs (at least two prescriptions for a type of medication in one year).
  Hazard ratios (HRs), with 95% confidence intervals, will be obtained to compare risk of diagnosis with a general medical condition in those with previous mental disorders, compared to those without. All persons, sex-specific and lagged (accounting for time since mental disorder diagnosis) HRs will be obtained. Additionally absolute risks will be calculated.
Musculoskeletal System general medical conditions | Diagnosed during the study period (2000-2016), after at least 1 year of age
  These will be ascertained using the following criteria:
  Diagnosis in the Danish National Patient Register or death in the Cause of Death register, for at least one of the following diseases: connective tissue disorders, osteoporosis.
  Records in the Danish National Prescription Register for at least one of the following types of medications: osteoporosis drugs (at least two prescriptions for a type of medication in one year) or repeated prescriptions for analgesics (at least four times in one year).
  Hazard ratios (HRs), with 95% confidence intervals, will be obtained to compare risk of diagnosis with a general medical condition in those with previous mental disorders, compared to those without. All persons, sex-specific and lagged (accounting for time since mental disorder diagnosis) HRs will be obtained. Additionally absolute risks will be calculated.
Risk of Neurological System general medical conditions | Diagnosed during the study period (2000-2016), after at least 1 year of age
  These will be ascertained using the following criteria:
  Diagnosis in the Danish National Patient Register or death in the Cause of Death register, for at least one of the following diseases: vision problems, hearing problems, migraine, epilepsy*, Parkinson's Disease, multiple sclerosis, neuropathies.
  Records in the Danish National Prescription Register for at least one of the following types of medications: specific anti-migraine drugs, antiepileptic drugs* (at least two prescriptions for a type of medication in one year)
  *Both a diagnosis of epilepsy AND two prescriptions of an antiepileptic drug in one year are required.
  Hazard ratios (HRs), with 95% confidence intervals, will be obtained to compare risk of diagnosis with a general medical condition in those with previous mental disorders, compared to those without. All persons, sex-specific and lagged (accounting for time since mental disorder diagnosis) HRs will be obtained. Additionally absolute risks will be calculated.
Risk of Hematological System general medical conditions | Diagnosed during the study period (2000-2016), after at least 1 year of age
  These will be ascertained using the following criteria:
  Diagnosis in the Danish National Patient Register or death in the Cause of Death register, for at least one of the following diseases: HIV/AIDS, anemias.
  Hazard ratios (HRs), with 95% confidence intervals, will be obtained to compare risk of diagnosis with a general medical condition in those with previous mental disorders, compared to those without. All persons, sex-specific and lagged (accounting for time since mental disorder diagnosis) HRs will be obtained. Additionally absolute risks will be calculated.
Risk of Cancers | Diagnosed during the study period (2000-2016), after at least 1 year of age
  These will be ascertained using the following criteria:
  Cancer diagnosis in the Danish National Patient Register or death in the Cause of Death register.
  Hazard ratios (HRs), with 95% confidence intervals, will be obtained to compare risk of diagnosis with a general medical condition in those with previous mental disorders, compared to those without. All persons, sex-specific and lagged (accounting for time since mental disorder diagnosis) HRs will be obtained. Additionally absolute risks will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: John J McGrath, MD, PhD, Principal Investigator — National Centre for Register-Based Research, Aarhus University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Momen NC, Plana-Ripoll O, Agerbo E, Benros ME, Borglum AD, Christensen MK, Dalsgaard S, Degenhardt L, de Jonge P, Debost JPG, Fenger-Gron M, Gunn JM, Iburg KM, Kessing LV, Kessler RC, Laursen TM, Lim CCW, Mors O, Mortensen PB, Musliner KL, Nordentoft M, Pedersen CB, Petersen LV, Ribe AR, Roest AM, Saha S, Schork AJ, Scott KM, Sievert C, Sorensen HJ, Stedman TJ, Vestergaard M, Vilhjalmsson B, Werge T, Weye N, Whiteford HA, Prior A, McGrath JJ. Association between Mental Disorders and Subsequent Medical Conditions. N Engl J Med. 2020 Apr 30;382(18):1721-1731. doi: 10.1056/NEJMoa1915784. PMID 32348643